CLINICAL TRIAL: NCT02635399
Title: Impact of Additional DJ (Duodenojejunostomy)-Pexy on Reduction in Delayed Gastric Emptying Following Pylorus-preserving Pancreaticoduodenectomy: A Prospective, Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2015-0969
Record Dates: First submitted 2015-12-15; First posted 2015-12-18 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Delayed Gastric Emptying
Keywords: pancreaticoduodenectomy, delayed gastric emptying, duodenojejunopexy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional group (Placebo Comparator): Conventional PPPD
  Interventions: Procedure: PPPD (pylorus-preserving pancreaticoduodenectomy)
- DJ-pexy group (Experimental): PPPD with additional DJ-pexy to anchor DJ to transverse colon
  Interventions: Procedure: PPPD (pylorus-preserving pancreaticoduodenectomy) with DJ-pexy

INTERVENTIONS:
Procedure: PPPD (pylorus-preserving pancreaticoduodenectomy) — pylorus-preserving pancreaticoduodenectomy is done in a conventional method. Additional DJ-pexy is performed for experimental group. DJ-pexy is performed by anchoring DJ site to transverse colon so that DJ is fixed to its original position.
  Arms: conventional group
Procedure: PPPD (pylorus-preserving pancreaticoduodenectomy) with DJ-pexy — pylorus-preserving pancreaticoduodenectomy is done in a conventional method. Additional DJ-pexy is performed for experimental group. DJ-pexy is performed by anchoring DJ site to transverse colon so that DJ is fixed to its original position.
  Arms: DJ-pexy group

SUMMARY:
Surgical resection in periampullary cancer using pancreaticoduodenectomy is the most important modality in the treatment. In the past, pancreaticoduodenectomy was associated with high morbidity and mortality. However, with the advances in techniques, including perioperative patient management, development of antibiotics, diagnostic radiology, and interventional treatments, pancreaticoduodenectomy is now considered a safe and feasible operation. Postoperative complication rates are reported to be in 10 to 20% in experienced hospitals and operation related mortality is at about 1%. Therefore, surgical treatment for periampullary cancer is actively considered.

However, postoperative complications, such as postoperative pancreatic fistula, (POPF) delayed gastric emptying, intraabdominal abscess, and postoperative bleeding, are still serious complications. Among these complications, delayed gastric emptying is considered less critical. However, delayed gastric emptying (DGE) can cause poor oral intake, which in turn, may lead to delay in recovery of postoperative nutritional state and in severe cases, requires insertion of levine tube and long-term fasting.

There have been many hypotheses for cause of DGE after pancreaticoduodenectomy, but definite cause have not been discovered yet. With the introduction of pylorus-preserving pancreaticoduodenectomy (PPPD), incidences of DGE were initially reported to have increased. However, results of most randomized comparative studies had concluded that PPPD and PD have no significance in occurence of DGE.

One hypothesis for cause of DGE we present here has to do with anatomic positioning of anastomosis site, especially pancreatojejunostomy (PJ) and duodenojejunostomy (DJ), after PPPD. Reconstruction after PPPD positions PJ and DJ close to each other. PJ site is often associated with one of postoperative complications, POPF. POPF may create inflammation around PJ site and pancreatitis, which may lead to severe adhesion around PJ as a secondary change. This adhesion and inflammation may cause DJ, which is located near PJ, to be pulled towards PJ site. When DJ is pulled towards PJ site, distal DJ site can become angulated and gastric contents may not beadle to pass easily. Gastric contents may be stagnated in stomach and thereby causing DGE. Therefore, in this study, we will fixate DJ on transverse colon using sutures, and prevent possibility of angulation of DJ. This additional procedure may reduce occurence of DGE.

ELIGIBILITY:
Inclusion Criteria:

* All periampullary pathologic conditions that require PPPD
* Age ≥20 and ≤80
* General performance status: the Karnofsky score> 70% or ECOG 0-1

Exclusion Criteria:

* Unresectable or locally advanced, metastatic case
* patients who do not want surgery
* ASA (American society of anesthesiologists' physical status classification) score: ≥3
* patients with drug or alcohol addiction
* patients showing low compliance
* patients who not want to involve the clinical trial
* patients who are unable to read or understand the informed consent, sign a consent form (eg, mental retardation, blindness, illiteracy, foreign, etc.)
* pylorus can not be preserved
* Patients undergoing laparoscopic PPPD
* Additional resection of adjacent organs or vascular resection was performed
* Previous history of open surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of clinically relevant DGE | With the first 30days after surgery
  DGE is defined by International Study Group of Pancreatic Surgery consensus definition. Clinically relevant grade B or C will be recorded and occurrence rate of DGE between the arms will be compared.

SECONDARY OUTCOMES:
Risk factors influencing DGE | Within the first 30 days after surgery
  Preoperative, intraoperative, and postoperative variables will analyzed statistically between the arms

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AS, Hawkins WG, Linehan DC, Strasberg SM. A technique of gastrojejunostomy to reduce delayed gastric emptying after pancreatoduodenectomy. J Gastrointest Surg. 2011 Aug;15(8):1468-71. doi: 10.1007/s11605-011-1471-4. Epub 2011 Feb 24. PMID 21347870